CLINICAL TRIAL: NCT01304953
Title: Tropisetron on Postoperative Pain in Women After Gynaecological Laparoscopy
Brief Title: Tropisetron on Postoperative Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Prof. Yuke Tian, Department of Anesthesiology, Tongji Hospital, Tongji medical college, Huazhong University of science and Technology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TJHMZK11001
Record Dates: First submitted 2011-02-25; First posted 2011-02-28 (Estimated); Last update posted 2011-02-28 (Estimated); Status verified 2011-02

CONDITIONS: Pain, Postoperative
Keywords: General anaesthetics; gynaecological laparoscopy; anaesthetic i.v.; propofol; anaesthetic volatile; evoflurane; antiemetics; reopisetron; postoperative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- P+P (Placebo Comparator)
  Interventions: Drug: Group P+P
- P+T (Experimental)
  Interventions: Drug: Group P+T
- S+P (Placebo Comparator)
  Interventions: Drug: Group S+P
- S+T (Experimental)
  Interventions: Drug: Group S+T

INTERVENTIONS:
Drug: Group P+P — In this arm, anaesthesia was maintained with propofol and remifentanil (0.1 μg kg-1 min-1), and primary anaesthetic namely propofol was titrated to maintain intraoperative BIS values between 45 and 55. If the patient did not respond to increases in the level of primary anaesthetic, additional doses of remifentanil up to 0.2 μg kg-1 min-1 were permitted to provide a more cardio-stable anaesthesia.
  Patients in this arms received saline placebo i.v. after the induction of anaesthesia.
  Arms: P+P
Drug: Group P+T — In this arm, anaesthesia was maintained with propofol and remifentanil (0.1 μg kg-1 min-1), and primary anaesthetic namely propofol was titrated to maintain intraoperative BIS values between 45 and 55. If the patient did not respond to increases in the level of primary anaesthetic, additional doses of remifentanil up to 0.2 μg kg-1 min-1 were permitted to provide a more cardio-stable anaesthesia.
  Patients in this arms received tropisetron 2 mg i.v. after the induction of anaesthesia.
  Arms: P+T
Drug: Group S+P — In this arm, anesthesia was maintained by sevoflurane and remifentanil (0.1 μg kg-1 min-1), and primary anaesthetic namely sevoflurane was titrated to maintain intraoperative BIS values between 45 and 55. If the patient did not respond to increases in the level of primary anaesthetic, additional doses of remifentanil up to 0.2 μg kg-1 min-1 were permitted to provide a more cardio-stable anaesthesia.
  Patients in this arms received saline placebo i.v. after the induction of anaesthesia.
  Arms: S+P
Drug: Group S+T — In this arm, anesthesia was maintained by sevoflurane and remifentanil (0.1 μg kg-1 min-1), and primary anaesthetic namely sevoflurane was titrated to maintain intraoperative BIS values between 45 and 55. If the patient did not respond to increases in the level of primary anaesthetic, additional doses of remifentanil up to 0.2 μg kg-1 min-1 were permitted to provide a more cardio-stable anaesthesia.
  Patients in this arms received tropisetron 2 mg i.v. after the induction of anaesthesia.
  Arms: S+T

SUMMARY:
The role of 5-HT3A receptors in nociceptive processing has been demonstrated in several animal models. However, studies in human volunteers have not been reported except for one recent study suggesting that ondansetron could alleviate propofol-induced nociception. Previous studies demonstrated that patients anaesthetized with sevoflurane have more pain than those anaesthetized with propofol. And we further posit that the difference is due to the nociceptive processing induced by the action of 5-HT3A receptors.

In this prospective, randomized, double-blind, placebo-controlled study, we assessed the analgesic action of a 5-HT3A receptor antagonist (tropisetron) in women after gynaecological laparoscopy under general anaesthesia maintained with either sevoflurane or propofol.

ELIGIBILITY:
Inclusion Criteria:

* female patients
* American Society of Anaesthesiologists Physical Status (ASA-PS) I or II
* undergoing selective gynaecological laparoscopies for infertilities

Exclusion Criteria:

* aged under 18 years old
* body mass index (BMI) > 30
* history of cardiovascular disease
* history of respiratory disease
* history of neurologic disease
* history of chronic antidepressants
* history of anxiolytics
* history of chronic analgesics intake
* participating in other studies

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 296 (Actual)
Dates: Start 2010-01; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Postoperative pain at rest | At 0.5 postoperative hour
  The primary outcome was the postoperative pain at rest assessed by numeric analog score (NAS, where 0 indicates no pain, and 10 indicates the most severe pain) immediately after awaking.

SECONDARY OUTCOMES:
Postoperative pain at rest | At 2,4,6,8,10,12,14,16,18,20,22,24 postoperative hours
  The patients were instructed to give the number that represented the pain level at rest soon after awakening, the first 30 min postoperatively, and every 2 hours within the first 24 postoperative hours.
Intraoperative hemodynamic values | At 5, 10,15,20,25,30 min after induction and 30, 25, 20, 15,10,5 min before last suture
  Heart rate and mean arterial pressure (MAP) every 5 min within 30 min after induction and 30 min before last suture
Postoperative shivering | At 24 hour postoperativelly
  The incidence of shiver within 24 h was recorded.
The incidence of postoperative nausea and vomiting (PONV) | At 24 hour postoperativelly
  The incidence of postoperative nausea and vomiting (PONV) was recorded at 24 h after surgery.
Quality of Recovery Score 40 | At 24 postoperative hour
  Quality of Recovery Score 40 was determined at 24 hours postoperativelly

CONTACTS AND LOCATIONS:
Overall Officials: Wei Mei, Study Director — Department of Anaesthesiology, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, 1095 Jiefang Avenue, Wuhan 430030, China; Yuke Tian, MD., Study Chair — Department of Anaesthesiology, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, 1095 Jiefang Avenue, Wuhan 430030, China
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China